CLINICAL TRIAL: NCT04075110
Title: Investigation the Safety and Efficacy of The Antileukotriene Agents, Montelukast, as Adjuvant Therapy in Obese Patients With Type 2 Diabetes Mellitus: A Randomized, Controlled Trial
Brief Title: Investigation the Safety and Efficacy of The Antileukotriene Agents, Montelukast, as Adjuvant Therapy in Obese Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Sadat City University (Other)
Responsible Party: Principal Investigator, Mahmoud Samy Abdallah, Lecturer of Clinical Pharmacy, PhD., Sadat City University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7-2021INTM1
Record Dates: First submitted 2019-08-28; First posted 2019-08-30 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: Obesity; Endocrine; Diabetes Type 2
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2 | interventions — montelukast

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control group (Placebo Comparator): 50 patients will receive metformin up to 2000mg/daily (Control group)
  Interventions: Drug: Placebo
- Montelukast group (Experimental): 50 patients will receive a combination of metformin up to 2000 mg/daily and montelukast (10 mg /day).
  Interventions: Drug: Montelukast 10mg

INTERVENTIONS:
Drug: Montelukast 10mg — Montelukast is an orally dosed drug (available as a chewable tablet) which is FDA-approved for the treatment of chronic asthma and prophylaxis and the prevention of exercise-induced bronchoconstriction. It is also approved for the relief of symptoms of both seasonal and perennial allergic rhinitis.
  Arms: Montelukast group
Drug: Placebo — Placebo tablet once daily
  Arms: Control group

SUMMARY:
The aim of the current study is to evaluate the safety and efficacy of Montelukast in treatment of obese patients with type 2 diabetes (T2DM).

ELIGIBILITY:
Inclusion Criteria:

- type 2 diabetic patients who had body mass index (BMI) ≥ 30 kg/m2 , were treated with metformin alone and had ages ranging from 18 to 60 years.

Exclusion Criteria:

* patients who had any other inflammatory disease
* patients with cardiovascular,
* patients with asthma
* patients with severe hepatic
* patients with renal disease,
* patients with epilepsy
* pregnant or lactating females.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2023-04-10 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c | From baseline to 12 weeks
  HbA1c
Percent change in body weight | From baseline to 12 weeks
  Body Weight
BMI | From baseline to 12 weeks
  body mass index
Visceral Adiposity Index | From baseline to 12 weeks
  visceral fat

SECONDARY OUTCOMES:
Adiponectin | At baseline to 12 weeks
  Serum level of adiponectin
TNF-α | At baseline to 12 weeks
  Serum level of Tumor necrosis factor alpha (TNF-α)
IL-6 | At baseline to 12 weeks
  Serum level of interleukin-6 (IL-6)
leukotriene B4 | At baseline to 12 weeks
  Serum level of leukotriene B4 (LTB4)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Shebin Elkom, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Derived] El-Khateeb E, El-Berri EI, Mosalam EM, Nooh MZ, Abdelsattar S, Alghamdi AM, Alrubia S, Abdallah MS. Evaluating the safety and efficacy of the leukotriene receptor antagonist montelukast as adjuvant therapy in obese patients with type 2 diabetes mellitus: A double-blind, randomized, placebo-controlled trial. Front Pharmacol. 2023 Apr 11;14:1153653. doi: 10.3389/fphar.2023.1153653. eCollection 2023. PMID 37113754